CLINICAL TRIAL: NCT03832556
Title: Preoperative Evaluation of Neurogenic Myositis Ossificans or Neurogenic Para-osteo-arthritis: Comparison Between Computed Tomography and Magnetic Resonance Imaging in Preoperative Evaluation
Brief Title: Comparison Between CT and MRI in Preoperative Evaluation of Neurogenic Myositis Ossificans or Neurogenic Para-osteo-arthritis
Acronym: MON-IRM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 2018-A02783-52
Record Dates: First submitted 2019-01-25; First posted 2019-02-06 (Actual); Last update posted 2023-03-16 (Actual); Status verified 2023-03

CONDITIONS: Neurogenic Myositis Ossificans; Neurogenic Para-osteo-arthritis
Keywords: neurogenic myositis ossificans; para-osteo-arthropathy; preoperative evaluation; CT scan; MRI

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Preoperative evaluation: CT + MRI (Experimental): Preoperative evaluation by 2 examinations: CT scan and MRI.
  * CT scan with biphasic injection of contrast product;
  * MRI with injection of contrast.
  Interventions: Other: CT scan; Other: MRI examination

INTERVENTIONS:
Other: CT scan — CT scan with biphasic injection of contrast product
Other: MRI examination — MRI with injection of contrast

SUMMARY:
The principal objective of the study is to compare between CT and MRI diagnostic performance (sensibility and specificity) in the preoperative assessment of neurogenic para-osteo-arthritis.

The second objectives of the study are:

* besides the diagnostic performance (sensibility and specificity), to evaluate the imaging par MRI in visual and descriptive manner heterotopic ossification and connection with vascular and nervous structures.
* to study the concordance (two by two) of results of preoperative obtained by MRI and by CT and operative reports.
* to study the characteristics of patients with discordant findings (two by two) by MRI, CT scan and operative report.

DETAILED DESCRIPTION:
This is a study on diagnostic performance, non randomized, versus Gold standard (a prospective multicentric cohort).

All eligible patients will be proposed consecutively to participate to the study, to undergo preoperative CT scan and MRI examination as usual procedure. The only additional action in this study will be a neurography sequence of type fluorescence subtraction imaging (FSI) during MRI, permitting to obtain more details in visualization of nerve structure and their relations of the ossifications.

The enrollment visit will performed by neuro-orthopaedic surgeon during preoperative consultation.

The follow-up visit will be an usual post-operative visit, non-specific for the study.

The duration for each participant will compound 1 month (the duration between preoperative imaging and surgical resection) added by up to two months of post-operative follow-up.

ELIGIBILITY:
Inclusion Criteria:

* Adult patient with neurogenic para-osteo-arthropathy resulted by prior central nervous system, cerebral or medullar damage
* Deformation with limitation of articular amplitude which could result limitation in rehabilitation care
* An indication of partial or total surgical excision of heterotopic ossification
* Indication of pre-operative assessment by CT scan and MRI, with contrast product injection
* Signed consent of patient obtained after clear and relevant informations given by physician
* Patient covered by social security

Exclusion Criteria:

* Contraindications to an MRI examination: cardiac stimulator, metallic intraocular foreign bodies...
* Contraindications to CT scan
* Contraindications to contrast injection product, such as iodinated or gadolinium-based contrast media
* Impractical venous access
* Severe deformation resulting impossibility to positioning for MRI examination or CT scan
* Patient can not give consent
* Participation to another interventional study
* Patient under guardianship

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2019-04-30 (Actual); Primary Completion 2023-02-07 (Actual); Study Completion 2023-02-07 (Actual)

PRIMARY OUTCOMES:
Analysis and comparison of accurate topography of heterotopic ossification on the CT and the MRI | through study completion, an average of 2 year
  Comparison of preoperative diagnostic performances of CT scan and MRI, based on analysis of topography of heterotopic ossification.
  On each CT and MRI exam, analysis of accurate topography of heterotopic ossifications relative to the bones, the number of fragments, their relationships with the articular capsule, their mineralization, and the mineralization of the underlying bone.
Analysis and comparison of reporting arterial and venous anatomy | through study completion, an average of 2 year
  Comparison of preoperative diagnostic performances of CT scan and MRI, based on analysis of reporting arterial and venous anatomy.
  On each CT and MRI exam, analysis of vascular (arterial and veinous) relations with the heterotopic ossifications, in the case of contact specify the existence of a gutter or a tunnel, and the vessels permeability or occlusion.
Analysis and comparison of reporting nervous structures | through study completion, an average of 2 year
  Comparison of preoperative diagnostic performances of CT scan and MRI, based on analysis of reporting nervous structures.
  On each CT and MRI exam, analysis of nervous structures relations with the heterotopic ossifications, in the case of contact specify the existence of a gutter or a tunnel, and the the existence of suffering nerve or denervation signs.

SECONDARY OUTCOMES:
Performances of MRI for diagnosis of arterial-venous | through study completion, an average of 2 year
  Performances of MRI for diagnosis of arterial-venous relation (gutter, stenosis, thrombosis or vascular occlusion, collateral circulation...)
Performances of MRI for diagnosis of nervous structures (nerve's location, nerve signal anomalies, signs of suffering and denervation...) | through study completion, an average of 2 year
Rate of incidence of adverse event during surgical operation | through study completion, an average of 2 year
  The rate of incidence of adverse event during surgical procedure will be calculated.
Concordance correlation coefficient | through study completion, an average of 2 year
  Concordance correlation coefficient two by two (Gwet concordance coefficient for binary qualitative variables; and W of Kendal concordance coefficient for ordinal qualitative variables or quantitative variables) between results of preoperative MRI and CT and operative report describing arterial-venous relation, and nervous structures.
Characteristic of patients with discordant results | through study completion, an average of 2 year
  Identify all discordances between CT or MRI and the surgery findings, about topography of heterotopic ossification, vascular relations and nervous structures relations.
  Analysis of characteristics of patients with discordant results between preoperative MRI resluts or preoperative CT results relative to the operative report.

CONTACTS AND LOCATIONS:
Overall Officials: Robert Carlier, MD, PhD, Principal Investigator — Service d'Imagerie médicale, Hôpital Raymond Poincaré, Garches; Raphaël AMAR, Resident, Study Director — Service d'Imagerie médicale, Hôpital Raymond Poincaré, Garches
Locations (1):
- Service d'Imagerie médicale, Hôpital Raymond Poincaré, Garches, Hauts-de-Seine, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Amar R, Thiry T, Salga M, Safa D, Chetrit A, Gatin L, Carlier RY. Comparison of magnetic resonance imaging and computed tomography for bone assessment of neurogenic heterotopic ossification of the hip: a preliminary study. J Orthop Surg Res. 2021 Dec 20;16(1):725. doi: 10.1186/s13018-021-02869-6. PMID 34930354